CLINICAL TRIAL: NCT02914509
Title: A Prospective, Multicenter, Randomized, Parallel-Arm, Double Masked, Vehicle Controlled Phase 3A Study Evaluating the Safety and Efficacy of OTX-TP in the Treatment of Subjects With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Phase 3 Study Evaluating Safety and Efficacy of OTX-TP in Subjects With OAG or OHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-16-002
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- OTX-TP (sustained release travoprost) Intracanalicular Depot (Experimental): OTX-TP (sustained release travoprost) Intracanalicular Depot
  Interventions: Drug: Travoprost
- PV (Placebo Vehicle) Intracanalicular Depot (Placebo Comparator): PV (Placebo Vehicle) Intracanalicular Depot
  Interventions: Other: Placebo Vehicle

INTERVENTIONS:
Drug: Travoprost
  Arms: OTX-TP (sustained release travoprost) Intracanalicular Depot
Other: Placebo Vehicle
  Arms: PV (Placebo Vehicle) Intracanalicular Depot

SUMMARY:
The objective of the study is to evaluate evaluate the safety and IOP lowering efficacy of OTX-TP, a sustained release travoprost drug product, placed in the canaliculus of the eyelid in the treatment of subjects with open-angle glaucoma or ocular hypertension

DETAILED DESCRIPTION:
This was a prospective, multicenter, randomized, parallel-arm, double masked, placebo vehicle (PV) controlled study conducted to evaluate the safety and IOP-lowering efficacy of OTX-TP, a sustained release drug product placed in the canaliculus of the eyelid in subjects with open-angle glaucoma or ocular hypertension. A total of up to 550 subjects (1100 eyes) with a clinical diagnosis of open-angle glaucoma or ocular hypertension in both eyes received either OTX-TP or PV to evaluate the safety and efficacy of OTX-TP.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ocular hypertension with an open angle of Schaffer Grade 3 or greater or open-angle glaucoma without pseudoexfoliation or pigment dispersion or evidence of traumatic angle recession
* IOP is currently controlled as assessed by the Investigator

Exclusion Criteria:

* Punctum size smaller than 0.4 mm or greater than 0.9 mm in either eye as measured using a standard punctum gauge
* A history of an inadequate response or no response to topical prostaglandin
* Known or suspected allergy and/or hypersensitivity to travoprost or any prostaglandin, fluorescein, or to any component of the study products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Artesia, California
  - Colorado Springs, Colorado
  - Lakeland, Florida
  - Morrow, Georgia
  - Shawnee Mission, Kansas
  - Des Peres, Missouri
  - Rochester, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OTX-TP: Three forty eight (348) subjects were randomized to OTX-TP
- Placebo Vehicle (PV): Two hundred seventeen (217) subjects were randomized to the PV.
Period: Overall Study
Arm/Group | OTX-TP | Placebo Vehicle (PV)
Started | 348 | 217
Completed | 343 | 211
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- OTX-TP (Sustained Release Travoprost) Intracanalicular Depot: Three hundred forty eight (348) subjects were randomized to OTX-TP
- Total: Total of all reporting groups
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV) | Total
Number analyzed (Participants) | 348 | 217 | 565
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 160 | 91 | 251
  >=65 years | 188 | 126 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 65 (11) | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 135 | 320
  Male | 163 | 82 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 247 | 159 | 406
  African American | 84 | 48 | 132
  Other | 17 | 10 | 27
Region of Enrollment [Number; unit: participants]
  United States | 348 | 217 | 565

OUTCOME MEASURES:

1. Primary Outcome: Mean IOP
Time Frame: Mean IOP at 8AM, 10AM, and 4PM at the 2 Week Visit
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV)
Number analyzed (Participants) | 343 | 211
mmHg
  8AM | 21 (0.2) | 22.9 (0.2)
  10AM | 20.2 (0.2) | 21.9 (0.2)
  4PM | 19.5 (0.2) | 21.5 (0.2)

2. Primary Outcome: Mean IOP
Time Frame: Mean IOP at 8AM, 10AM, and 4PM at the 6 Week Visit
Measure: Mean (Standard Error); unit: mmHg
Groups:
- OTX-TP (Sustained Release Travoprost) Intracanalicular Depot: Three hundred forty eight (343) subjects were randomized to OTX-TP
- Placebo Vehicle (PV): Two hundred seventeen (211) subjects were randomized to the PV.
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV)
Number analyzed (Participants) | 343 | 211
mmHg
  8AM | 21.9 (0.2) | 26.9 (0.3)
  10AM | 25.1 (0.2) | 25 (0.2)
  4PM | 24.8 (0.2) | 24.6 (0.2)

3. Primary Outcome: Mean IOP
Time Frame: Mean IOP at 8AM, 10AM, and 4PM at the 12 Week Visit
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV)
Number analyzed (Participants) | 343 | 211
mmHg
  8AM | 22.8 (0.2) | 23.2 (0.3)
  10AM | 21.7 (0.2) | 22.5 (0.2)
  4PM | 21.4 (0.2) | 22.1 (0.2)

4. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events
Description: Number of Participants with Serious Adverse Events
Time Frame: Through study completion, an average of 23 months
Measure: Count of Participants; unit: Participants
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV)
Number analyzed (Participants) | 348 | 217
Participants | 7 | 6

ADVERSE EVENTS:
Time Frame: through study duration, an average of 23 months
Arm/Group | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot | Placebo Vehicle (PV)
All-Cause Mortality (participants affected / at risk) | 1/348 | 0/217
Serious Adverse Events (participants affected / at risk) | 7/348 | 6/217
Other Adverse Events (participants affected / at risk) | 132/348 | 65/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot (N=348) | Placebo Vehicle (PV) (N=217)
Serious Adverse Event (Nervous system disorders) | 2 | 0
Serious Adverse Event (Infections and infestations) | 1 | 2
Serious Adverse Event (Cardiac disorders) | 1 | 1
Serious Adverse Event (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Serious Adverse Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Serious Adverse Event (Vascular disorders) | 1 | 0
Serious Adverse Event (Skin and subcutaneous tissue disorders) | 1 | 0
Serious Adverse Events (Ear and labyrinth disorders) | 0 | 1
Serious Adverse Event (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTX-TP (Sustained Release Travoprost) Intracanalicular Depot (N=348) | Placebo Vehicle (PV) (N=217)
Adverse Event (General disorders) | 132 | 65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02914509/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02914509/SAP_001.pdf